CLINICAL TRIAL: NCT05237687
Title: Sirolimus in Older Adults- Randomized Trial Assessing the Improvement in Phenotypic/Functional Biomarkers of Aging
Brief Title: The Role of Sirolimus in Preventing Functional Decline in Older Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Irina Timofte (Other)
Responsible Party: Sponsor-Investigator, Irina Timofte, Associate Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2023-0909
Record Dates: First submitted 2022-01-19; First posted 2022-02-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Aging
Keywords: aging; sirolimus; prevention
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients will be randomized using age-based randomization to initial treatment with 0.5 mg sirolimus p.o. (orally) everyday vs standard of care. The medications would be dispensed from UT Southwestern Medical Center. To ensure patent's safety, all patients will be closely monitored. We will start with a 0.5 mg tablet- the smallest sirolimus dose available. Sirolimus level will be checked weekly in the first month to ensure we maintain a low goal (5-7) that will decrease the risk of developing side effects. In order to monitor study drug compliance, we will ask the patient to keep a pill diary. After the first month, the patient will have monthly blood work and monthly phone call to enquire about potential side effects. The patients will be followed in clinic in person every 3 months. Functional assessment will be obtained at baseline, 3 months 6 months 9 months and 1 year follow up. Completion of the 1-year treatment period will be followed by a follow-up phone call 1 month later.
  Interventions: Drug: Sirolimus
- Control (No Intervention): Interventions: standard of care Patients are not going to receive any additional intervention.

INTERVENTIONS:
Drug: Sirolimus — Patients will be randomly assigned to sirolimus or standard of care
  Arms: Intervention

SUMMARY:
Aging is associated with progressive impairment of tissue and organ function, resulting in increased susceptibility to chronic disease, frailty and disability. Currently there are limited treatment options to alter this inevitable process. The proposed work has the potential to identify a new therapeutic intervention to decrease aging-related degenerative processes.

Rapamycin or sirolimus is a macrocyclic immunosuppressive drug that inhibits the mammalian target of rapamycin (mTOR). The mammalian target of rapamycin (mTOR) pathway is part of phosphoinositide 3-kinase (PI3K)/protein kinase B (AKT)/mammalian target of rapamycin (mTOR)-dependent pathway which is a fundamentally linked to cell metabolism, proliferation, differentiation, and survival. This pathway is altered in a variety of diseases, including cancers, immunosuppressed states, and fibroproliferative diseases. The mTOR kinase is considered one of the leading regulators of this pathway. Changes in mTOR signaling are closely associated with inflammation, cell growth and survival, leading to the development of chronic diseases. Recent evidence also suggests that mTOR inhibitors are promising modulators of the aging process by slowing the mechanisms of aging at the cellular level. There is a growing appreciation of the potential impact of sirolimus in slowing aging processes and in prolonging healthy lifespan.

The proposed study addresses critical gaps in our understanding of the safety and efficacy of sirolimus in delaying aging processes and is based on findings in animal studies and incidental clinical observations. The investigators will overcome potential biases with a randomized control trial. The proposed intervention study is intended to improve our insight into clinical outcomes leading to prevention of chronic diseases such as skin cancer and mortality. Our overarching hypothesis is that sirolimus is one of the first pharmacological agents that will impact the aging process and chronic disease development. Specifically, the investigators aim to investigate whether sirolimus can reduce the occurrence or increase in biomarkers of aging processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be adults 65-80 years
* Women who are postmenopausal* or status post-surgical sterilization only
* Competent to provide Informed Consent

Exclusion Criteria:

* Creatinine clearance <30 mL/min
* Underlying chronic liver disease
* Other investigational therapy received within 1 month prior to screening visit
* Pulmonary Arterial Hypertension (PAH), mean Pulmonary Arterial Presure(mPAP)>30 mm Hg
* Extrapulmonary physiological restriction (e.g. chest wall abnormality, large pleural effusion)
* Cardiovascular diseases, any of the following: Myocardial infarction within 6 months, planned coronary artery disease intervention , left ventricular EF <45%

  * History of haemorrhagic central nervous system (CNS) event within 1 year from screening visit.
  * Any of the following within 3 months of screening visit :Haemoptysis or haematuria;Active gastro-intestinal (GI) bleeding or GI - ulcers; Major injury or surgery
* History of thrombotic event (including, DVT, PE, stroke and transient ischemic attack) within 1 year from screening visit.
* Other disease that may interfere with testing procedures or in the judgment of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
* Planned major surgical procedures.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Concurrent active alcohol or drug abuse.
* Clinically significant cognitive impairment
* Functional impairment (defined by ADL status)
* Patients not able to understand or follow trial procedures

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Phenotypic/functional biomarkers of aging | 1 year
  Phenotypic biomarkers of aging will be measured by SASP (senescence-associated secretory phenotype) index score at 1 year follow-up when compared to elderly patients not receiving sirolimus.

SECONDARY OUTCOMES:
Phenotypic/functional biomarkers of aging | 1 year
  Phenotypic/functional biomarkers of aging will be measured by walking speed at 1 year follow-up when compared to elderly patients not receiving sirolimus.
Phenotypic/functional biomarkers of aging | 1 year
  Functional biomarkers of aging will be measured by chair stand at 1 year follow-up when compared to elderly patients not receiving sirolimus.
Phenotypic/functional biomarkers of aging | 1 year
  Functional biomarkers of aging will be measured by standing balance at 1 year follow-up when compared to elderly patients not receiving sirolimus.
Phenotypic/functional biomarkers of aging | 1 year
  Phenotypic/functional biomarkers of aging will be measured by body mass index at 1 year follow-up when compared to elderly patients not receiving sirolimus.
Feasibility of collecting the laboratory biomarkers and analyzing the data regarding annual rate of decline in functional biomarkers of aging | 1 year
  The feasibility of collecting the laboratory biomarkers and analyzing the data regarding annual rate of decline in functional biomarkers of aging measured by walking speed, chair stand, standing balance, grip strength, body mass index, waist circumference, and muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Timofte, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamming DW, Ye L, Sabatini DM, Baur JA. Rapalogs and mTOR inhibitors as anti-aging therapeutics. J Clin Invest. 2013 Mar;123(3):980-9. doi: 10.1172/JCI64099. Epub 2013 Mar 1. PMID 23454761
- [Background] Hsu HS, Liu CC, Lin JH, Hsu TW, Hsu JW, Su K, Hung SC. Involvement of ER stress, PI3K/AKT activation, and lung fibroblast proliferation in bleomycin-induced pulmonary fibrosis. Sci Rep. 2017 Oct 27;7(1):14272. doi: 10.1038/s41598-017-14612-5. PMID 29079731
- [Background] Lawrence J, Nho R. The Role of the Mammalian Target of Rapamycin (mTOR) in Pulmonary Fibrosis. Int J Mol Sci. 2018 Mar 8;19(3):778. doi: 10.3390/ijms19030778. PMID 29518028